CLINICAL TRIAL: NCT06041867
Title: Mushboost: Evaluating the Effect of Agaricus Bisporus Powder Intake on the Vaccination Response to an Influenza Vaccine
Brief Title: Agaricus Bisporus and Influenza Vaccination Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Scelta Mycofriends B.V. (Unknown); CNC Grondstoffen B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 23-026
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-02

CONDITIONS: Immune Response
Keywords: Agaricus bisporus; Immune system; Influenza vaccination; Mushroom
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Agaricus bisporus group (Experimental): Dietary supplement: 10 capsules containing 500 mg Agaricus bisporus powder each
  Interventions: Biological: Influenza vaccine; Dietary Supplement: Agaricus bisporus capsules
- Placebo group (Placebo Comparator): Dietary supplement: 10 placebo capsules, capsules that do not contain Agaricus bisporus powder
  Interventions: Biological: Influenza vaccine; Dietary Supplement: Control capsules

INTERVENTIONS:
Biological: Influenza vaccine — Single dose of the Influenza vaccine Participants have to wait until they are invited to receive the vaccine by the general practitioner; this study does not interfere with national planning of the vaccine
Dietary Supplement: Agaricus bisporus capsules — Participants have to consume 10 capsules per day containing 500 mg Agaricus bisporus powder each, corresponding to a total Agariicus bisporus powder intake of 5 g daily
  Arms: Agaricus bisporus group
Dietary Supplement: Control capsules — Participants have to consume 10 capsules per day containing 500 mg maltodextrin each, corresponding to a total maltodextrin intake of 5 g daily
  Arms: Placebo group

SUMMARY:
There are numerous in vitro and animal studies that suggested that mushrooms beneficially influence the immune system. We have recently shown that a wild isolate of the edible Agaricus bisporus mushroom had a clear effect on parameters reflecting a better function of the immune system, both in vitro and in vivo in animals. The question now is whether this efficacy can also be translated to humans. In humans, measuring the antibody response is the golden standard to evaluate immune function. If Agaricus bisporus powder indeed has beneficial effects on the immune system, people with overweight or obesity and higher age might benefit from consuming Agaricus bisporus powder prior to receiving the influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older during influenza season 2023/2024 (in line with RIVM guidelines)
* BMI between 20 and 35 kg/m2
* Willing to abstain from mushrooms other than the capsules containing a mushroom powder as provided by us during the study period.
* Willing to keep the intake of fish oil, Zinc, Selenium and (vitamin) supplements constant
* Willing to abstain from products / supplements enriched with Vitamin D
* Willing to abstain from products / supplements enriched with plant sterols or stanols
* Willing to abstain from products / supplements enriched with (β)glucans or fungi.
* Willing to abstain from products / supplements that are mentioned to "boost your immune system"
* Willing to abstain from (products enriched in) pre/pro-biotics
* Willing to abstain from products/supplements enriched with ergothioneine

Exclusion Criteria:

* Already received influenza vaccination in 2023
* Allergy to mushrooms
* Known allergic reaction to an active component or other components of the vaccine (e.g. Chicken Eggs)
* Having donated blood within one month prior to the start of the study, or planning to donate blood during the study
* Excessive alcohol use (>20 consumptions per week)
* Regular use of soft and/or hard drugs
* Using medication for diseases known to affect inflammation/immunity (e.g. inhaled corticosteroids and prednisone)

Min Age: 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Vaccine specific antibody titer | Time Frame: Differences in influenza specific antibody titers at any measured time point ((Day=0 (day before vaccination), weekly in the month after vaccination (week 1, week 2, week 3 and week 4 after vaccination))
  The response to the Influenza vaccine will be measured by quantifying the specific antibody titer

SECONDARY OUTCOMES:
Immune parameters (1) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Cytokine production by PBMCs after stimulation with antiCD3-antiCD28 antiCD28 antibodies using the TruCulture system
Immune parameters (2) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  hsCRP
Leukocyte count | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Number of leukocytes measured in EDTA plasma
Leukocyte differential count | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Number of subgroups of leukocytes measured in EDTA plasma
Fasted metabolism (1) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Serum non-cholesterol sterols and stanols
Fasted metabolism (2) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Serum lipid and lipoprotein profile
Fasted metabolism (3) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Plasma glucose
Fasted metabolism (4) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Ergothioneine
Fasted metabolism (5) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Glutathione
Fasted metabolism (6) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Malondialdehyde
Anthropometry (1) | Day - 1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Body weight
Anthropometry (2) | Day -1 (start study)
  Height
Anthropometry (3) | Day - 1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Waist circumference
Anthropometry (4) | Day - 1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Hip circumference
Anthropometry (5) | Day - 1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Waist-to-hip ratio
Diet | Day - 1 (start study), T=4 weeks after vaccination (end of study)
  Food frequency questionnaire is used to determine if the participants maintain their habitual diet and to determine if the participants do not consume mushrooms outside the intervention
Quality of life questionnaire | Day - 1 (start study), T=4 weeks after vaccination (end of study)
  Quality of life questionnaire is used to determine the participants overall wellbeing and quality of life
Diary outcomes (1) | Day - 1 (start study), T=4 weeks after vaccination (end of study)
  Adverse events as assessed by the diary
Diary outcomes (2) | Day - 1 (start study), T=4 weeks after vaccination (end of study)
  Medication intake as assessed by the diary

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No